CLINICAL TRIAL: NCT05142410
Title: A Retrospective Study Using Mass Spectrometry to Characterize Post-translational Modifications to Circulating Histones in Pregnant Women Developing Pre-eclampsia
Brief Title: Understanding Post-translational Modifications to Circulating Histones Via Mass Spectrometry in Pregnant Women Developing Pre-eclampsia: A Retrospective Study
Acronym: GHISPE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2021-1/SB01
Record Dates: First submitted 2021-11-18; First posted 2021-12-02 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Pregnancy Related; Pre-Eclampsia
Keywords: Pregnancy; Pre-eclampsia; Histones; Mass spectrometry; Neutrophils; Extracellular traps
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — This study is based on the mass spectrometric analysis of frozen plasma samples from patients included in the "GrossPath" cohort (BCR ID: 2014-A01120-47). The benefits will ultimately be a better understanding of the physiopathological mechanisms involved in the occurrence of this placental vascular pathology.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Plasma from women with normal pregnancies: Plasma collected from women with normal pregnancies will be analyzed by mass spectrometry
  Interventions: Diagnostic Test: Analysis of post-translational histone modifications via mass spectrometry
- Plasma from women with placenta-mediated complications: Plasma collected from women who developed preeclampsia during pregnancy will be analyzed by mass spectrometry
  Interventions: Diagnostic Test: Analysis of post-translational histone modifications via mass spectrometry

INTERVENTIONS:
Diagnostic Test: Analysis of post-translational histone modifications via mass spectrometry — During the "GrossHist" study (NCT04205383), only 3 post-translational histone modifications available in ELISA at the time were quantified thanks to a collaboration with the VOLITION™ company [Bouvier and Fortier et al. 2021]. The development of a new mass spectrometry approach based on nucleosome enrichment of plasma, developed by collaborators at VOLITION™, has made it possible to consider the description of all post-translational histone modifications (about 40 post-translational modifications involving histones H2A, H2B, H3 and H4).

SUMMARY:
This is a descriptive pilot study on a ready-constituted biobank (outside the Jardé Law). It is an ancillary study to the "GrossPath" cohort (RCB ID number: 2014-A01120-47).

Pregnancy generates an increased risk of thrombosis, and placenta-mediated diseases constitute a risk factor for cardiovascular pathologies responsible for significant maternal-fetal morbidity and mortality. Understanding and exploring the cellular and molecular mechanisms of dysfunctions of the vascular-placental interface could provide arguments to understand the systemic vascular risk, characterize it and finally detect it on the basis of new markers, thus opening the way for targeted preventive management to reinforce the general principles of precision medicine.

Netosis is a process of activation of neutrophils, which then generate filaments containing DNA, enzymes and extracellular histones. Netosis occurs in pregnancy and is increased in vascular-placental complications. It can be studied by measuring circulating histones, particularly the citrullinated histone H3. Levels of this modified histone H3, as well as those of two other modifications, have recently been shown to increase during pregnancy. These levels have also been shown to be even greater in pregnancy complications.

The aim of this study is to complete this mapping in order to obtain a precise signature for all post-translational histone modifications in normal pregnancies and pregnancies complicated by pre-eclampsia from the "GrossPath" cohort in order to propose new circulating biomarkers for placental vascular pathologies.

The post-translational histone modification profiles (mapping) of pregnant women with normal pregnancies will be compared with those developing pre-eclampsia.

ELIGIBILITY:
Inclusion Criteria:

* Not applicable as this study is on samples from a biobank. The inclusion criteria for the "GrossPath" cohort were:
* pregnant women followed at Nîmes University hospital for normal pregnancy or pregnancy with placental vascular pathology (pre-eclampsia and/or intra-uterine growth retardation).
* The patient must have given her free and informed consent and signed the consent form.
* The patient must be a member or beneficiary of a health insurance plan
* Only women are included
* Patients are at least 18 years old

Exclusion Criteria:

* Not applicable as this is a study on samples from a biobank. The non-inclusion criteria of the "GrossPath" cohort were :
* twin pregnancies.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The study is based on frozen plasma samples from pregnant women, taken at the time of them giving birth from among the 50 women who constituted the GrossPath cohort. Fourteen of these women had had normal pregnancies and fourteen had developed pre-eclampsia. Cases are matched on maternal age, clinical event (delivery) and gestational age will be included from the GrossPath cohort.
Study Population: The study is based on frozen plasma samples from pregnant women, taken at the time of them giving birth from among the 50 women who constituted the GrossPath cohort. Fourteen of these women had had normal pregnancies and fourteen had developed pre-eclampsia. Cases are matched on maternal age, clinical event (delivery) and gestational age will be included from the GrossPath cohort.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Presence of methylation in histone H2A in pregnant women with normal pregnancies | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry will be used to detect the presence or not of methylation in histone H2A and recorded as YES/NO.
Presence of methylation in histone H2A in pregnant women developing pre-eclampsia | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry will be used to detect the presence or not of methylation in histone H2A and recorded as YES/NO.
Presence of methylation in histone H2B in pregnant women with normal pregnancies | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry will be used to detect the presence or not of methylation in histone H2B and recorded as YES/NO.
Presence of methylation in histone H2B in pregnant women developing pre-eclampsia | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry will be used to detect the presence or not of methylation in histone H2B and recorded as YES/NO.
Presence of methylation in histone H3 in pregnant women with normal pregnancies | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry will be used to detect the presence or not of methylation in histone H3 and recorded as YES/NO.
Presence of methylation in histone H3 in pregnant women developing pre-eclampsia | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry will be used to detect the presence or not of methylation in histone H3 and recorded as YES/NO.
Presence of methylation in histone H4 in pregnant women with normal pregnancies | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry will be used to detect the presence or not of methylation in histone H4 and recorded as YES/NO.
Presence of methylation in histone H4 in pregnant women developing pre-eclampsia | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry will be used to detect the presence or not of methylation in histone H4 and recorded as YES/NO.
Presence of acetylation in histone H2A in pregnant women with normal pregnancies | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry will be used to detect the presence or not of acetylation in histone H2A and recorded as YES/NO.
Presence of acetylation in histone H2A in pregnant women developing pre-eclampsia | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry will be used to detect the presence or not of acetylation in histone H2A and recorded as YES/NO.
Presence of acetylation in histone H2B in pregnant women with normal pregnancies | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry will be used to detect the presence or not of acetylation in histone H2B and recorded as YES/NO.
Presence of acetylation in histone H2B in pregnant women developing pre-eclampsia | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry will be used to detect the presence or not of acetylation in histone H2B and recorded as YES/NO.
Presence of acetylation in histone H3 in pregnant women with normal pregnancies | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry will be used to detect the presence or not of acetylation in histone H3 and recorded as YES/NO.
Presence of acetylation in histone H3 in pregnant women developing pre-eclampsia | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry will be used to detect the presence or not of acetylation in histone H3 and recorded as YES/NO.
Presence of acetylation in histone H4 in pregnant women with normal pregnancies | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry will be used to detect the presence or not of acetylation in histone H4 and recorded as YES/NO.
Presence of acetylation in histone H4 in pregnant women developing pre-eclampsia | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry will be used to detect the presence or not of acetylation in histone H4 and recorded as YES/NO.
Presence of phosphorylation in histone H2A in pregnant women with normal pregnancies | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry will be used to detect the presence or not of phosphorylation in histone H2A and recorded as YES/NO.
Presence of phosphorylation in histone H2A in pregnant women developing pre-eclampsia | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry will be used to detect the presence or not of phosphorylation in histone H2A and recorded as YES/NO.
Presence of phosphorylation in histone H2B in pregnant women with normal pregnancies | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry will be used to detect the presence or not of phosphorylation in histone H2B and recorded as YES/NO.
Presence of phosphorylation in histone H2B in pregnant women developing pre-eclampsia | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry will be used to detect the presence or not of phosphorylation in histone H2B and recorded as YES/NO.
Presence of phosphorylation in histone H3 in pregnant women with normal pregnancies | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry will be used to detect the presence or not of phosphorylation in histone H3 and recorded as YES/NO.
Presence of phosphorylation in histone H3 in pregnant women developing pre-eclampsia | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry will be used to detect the presence or not of phosphorylation in histone H3 and recorded as YES/NO.
Presence of phosphorylation in histone H4 in pregnant women with normal pregnancies | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry will be used to detect the presence or not of phosphorylation in histone H4 and recorded as YES/NO.
Presence of phosphorylation in histone H4 in pregnant women developing pre-eclampsia | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry will be used to detect the presence or not of phosphorylation in histone H4 and recorded as YES/NO.
Presence of ubiquitination in histone H2A in pregnant women with normal pregnancies | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry will be used to detect the presence or not of ubiquitination in histone H2A and recorded as YES/NO.
Presence of ubiquitination in histone H2A in pregnant women developing pre-eclampsia | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry will be used to detect the presence or not of ubiquitination in histone H2A and recorded as YES/NO.
Presence of ubiquitination in histone H2B in pregnant women with normal pregnancies | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry will be used to detect the presence or not of ubiquitination in histone H2B and recorded as YES/NO.
Presence of ubiquitination in histone H2B in pregnant women developing pre-eclampsia | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry will be used to detect the presence or not of ubiquitination in histone H2B and recorded as YES/NO.
Presence of ubiquitination in histone H3 in pregnant women with normal pregnancies | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry will be used to detect the presence or not of ubiquitination in histone H3 and recorded as YES/NO.
Presence of ubiquitination in histone H3 in pregnant women developing pre-eclampsia | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry will be used to detect the presence or not of ubiquitination in histone H3 and recorded as YES/NO.
Presence of ubiquitination in histone H4 in pregnant women with normal pregnancies | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry will be used to detect the presence or not of ubiquitination in histone H4 and recorded as YES/NO.
Presence of ubiquitination in histone H4 in pregnant women developing pre-eclampsia | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry will be used to detect the presence or not of ubiquitination in histone H4 and recorded as YES/NO.
Presence of citrullination in histone H2A in pregnant women with normal pregnancies | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry will be used to detect the presence or not of citrullination in histone H2A and recorded as YES/NO.
Presence of citrullination in histone H2A in pregnant women developing pre-eclampsia | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry will be used to detect the presence or not of citrullination in histone H2A and recorded as YES/NO.
Presence of citrullination in histone H2B in pregnant women with normal pregnancies | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry will be used to detect the presence or not of citrullination in histone H2B and recorded as YES/NO.
Presence of citrullination in histone H2B in pregnant women developing pre-eclampsia | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry will be used to detect the presence or not of citrullination in histone H2B and recorded as YES/NO.
Presence of citrullination in histone H3 in pregnant women with normal pregnancies | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry will be used to detect the presence or not of citrullination in histone H3 and recorded as YES/NO.
Presence of citrullination in histone H3 in pregnant women developing pre-eclampsia | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry will be used to detect the presence or not of citrullination in histone H3 and recorded as YES/NO.
Presence of citrullination in histone H4 in pregnant women with normal pregnancies | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry will be used to detect the presence or not of citrullination in histone H4 and recorded as YES/NO.
Presence of citrullination in histone H4 in pregnant women developing pre-eclampsia | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry will be used to detect the presence or not of citrullination in histone H4 and recorded as YES/NO.

SECONDARY OUTCOMES:
Intensity of methylation in histone H2A in pregnant women with normal pregnancies | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry, quantitative
Intensity of methylation in histone H2A in pregnant women developing pre-eclampsia | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry, quantitative
Intensity of methylation in histone H2B in pregnant women with normal pregnancies | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry, quantitative
Intensity of methylation in histone H2B in pregnant women developing pre-eclampsia | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry, quantitative
Intensity of methylation in histone H3 in pregnant women with normal pregnancies | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry, quantitative
Intensity of methylation in histone H3 in pregnant women developing pre-eclampsia | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry, quantitative
Intensity of methylation in histone H4 in pregnant women with normal pregnancies | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry, quantitative
Intensity of methylation in histone H4 in pregnant women developing pre-eclampsia | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry, quantitative
Intensity of acetylation in histone H2A in pregnant women with normal pregnancies | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry, quantitative
Intensity of acetylation in histone H2A in pregnant women developing pre-eclampsia | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry, quantitative
Intensity of acetylation in histone H2B in pregnant women with normal pregnancies | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry, quantitative
Intensity of acetylation in histone H2B in pregnant women developing pre-eclampsia | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry, quantitative
Intensity of acetylation in histone H3 in pregnant women with normal pregnancies | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry, quantitative
Intensity of acetylation in histone H3 in pregnant women developing pre-eclampsia | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry, quantitative
Intensity of acetylation in histone H4 in pregnant women with normal pregnancies | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry, quantitative
Intensity of acetylation in histone H4 in pregnant women developing pre-eclampsia | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry, quantitative
Intensity of phosphorylation in histone H2A in pregnant women with normal pregnancies | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry, quantitative
Intensity of phosphorylation in histone H2A in pregnant women developing pre-eclampsia | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry, quantitative
Intensity of phosphorylation in histone H2B in pregnant women with normal pregnancies | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry, quantitative
Intensity of phosphorylation in histone H2B in pregnant women developing pre-eclampsia | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry, quantitative
Intensity of phosphorylation in histone H3 in pregnant women with normal pregnancies | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry, quantitative
Intensity of phosphorylation in histone H3 in pregnant women developing pre-eclampsia | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry, quantitative
Intensity of phosphorylation in histone H4 in pregnant women with normal pregnancies | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry, quantitative
Intensity of phosphorylation in histone H4 in pregnant women developing pre-eclampsia | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry, quantitative
Intensity of ubiquitination in histone H2A in pregnant women with normal pregnancies | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry, quantitative
Intensity of ubiquitination in histone H2A in pregnant women developing pre-eclampsia | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry, quantitative
Intensity of ubiquitination in histone H2B in pregnant women with normal pregnancies | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry, quantitative
Intensity of ubiquitination in histone H2B in pregnant women developing pre-eclampsia | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry, quantitative
Intensity of ubiquitination in histone H3 in pregnant women with normal pregnancies | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry, quantitative
Intensity of ubiquitination in histone H3 in pregnant women developing pre-eclampsia | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry, quantitative
Intensity of ubiquitination in histone H4 in pregnant women with normal pregnancies | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry, quantitative
Intensity of ubiquitination in histone H4 in pregnant women developing pre-eclampsia | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry, quantitative
Intensity of citrullination in histone H2A in pregnant women with normal pregnancies | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry, quantitative
Intensity of citrullination in histone H2A in pregnant women developing pre-eclampsia | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry, quantitative
Intensity of citrullination in histone H2B in pregnant women with normal pregnancies | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry, quantitative
Intensity of citrullination in histone H2B in pregnant women developing pre-eclampsia | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry, quantitative
Intensity of citrullination in histone H3 in pregnant women with normal pregnancies | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry, quantitative
Intensity of citrullination in histone H3 in pregnant women developing pre-eclampsia | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry, quantitative
Intensity of citrullination in histone H4 in pregnant women with normal pregnancies | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry, quantitative
Intensity of citrullination in histone H4 in pregnant women developing pre-eclampsia | At pregnancy term (max 41 weeks gestation)
  Mass spectrometry, quantitative
Presence of methylation in histone H2A in pregnant women developing pre-eclampsia before 34 weeks of pregnancy | Before 34 weeks of pregnancy
  YES/NO
Presence of methylation in histone H2A in pregnant women developing pre-eclampsia after 34 weeks of pregnancy | 34 to 41 weeks of pregnancy
  YES/NO
Presence of methylation in histone H2B in pregnant women developing pre-eclampsia before 34 weeks of pregnancy | Before 34 weeks of pregnancy
  YES/NO
Presence of methylation in histone H2B in pregnant women developing pre-eclampsia after 34 weeks of pregnancy | 34 to 41 weeks of pregnancy
  YES/NO
Presence of methylation in histone H3 in pregnant women developing pre-eclampsia before 34 weeks of pregnancy | Before 34 weeks of pregnancy
  YES/NO
Presence of methylation in histone H3 in pregnant women developing pre-eclampsia after 34 weeks of pregnancy | 34 to 41 weeks of pregnancy
  YES/NO
Presence of methylation in histone H4 in pregnant women developing pre-eclampsia before 34 weeks of pregnancy | Before 34 weeks of pregnancy
  YES/NO
Presence of methylation in histone H4 in pregnant women developing pre-eclampsia after 34 weeks of pregnancy | 34 to 41 weeks of pregnancy
  YES/NO
Presence of acetylation in histone H2A in pregnant women developing pre-eclampsia before 34 weeks of pregnancy | Before 34 weeks of pregnancy
  YES/NO
Presence of acetylation in histone H2A in pregnant women developing pre-eclampsia after 34 weeks of pregnancy | 34 to 41 of pregnancy
  YES/NO
Presence of acetylation in histone H2B in pregnant women developing pre-eclampsia before 34 weeks of pregnancy | Before 34 weeks of pregnancy
  YES/NO
Presence of acetylation in histone H2B in pregnant women developing pre-eclampsia after 34 weeks of pregnancy | 34 to 41 weeks of pregnancy
  YES/NO
Presence of acetylation in histone H3 in pregnant women developing pre-eclampsia before 34 weeks of pregnancy | Before 34 weeks of pregnancy
  YES/NO
Presence of acetylation in histone H3 in pregnant women developing pre-eclampsia after 34 weeks of pregnancy | After 34 weeks of pregnancy
  YES/NO
Presence of acetylation in histone H4 in pregnant women developing pre-eclampsia before 34 weeks of pregnancy | Before 34 weeks of pregnancy
  YES/NO
Presence of acetylation in histone H4 in pregnant women developing pre-eclampsia after 34 weeks of pregnancy | 34 to 41 weeks of pregnancy
  YES/NO
Presence of phosphorylation in histone H2A in pregnant women developing pre-eclampsia before 34 weeks of pregnancy | Before 34 weeks of pregnancy
  YES/NO
Presence of phosphorylation in histone H2A in pregnant women developing pre-eclampsia after 34 weeks of pregnancy | 34 to 41 weeks of pregnancy
  YES/NO
Presence of phosphorylation in histone H2B in pregnant women developing pre-eclampsia before 34 weeks of pregnancy | Before 34 weeks of pregnancy
  YES/NO
Presence of phosphorylation in histone H2B in pregnant women developing pre-eclampsia after 34 weeks of pregnancy | 34 to 41 weeks of pregnancy
  YES/NO
Presence of phosphorylation in histone H3 in pregnant women developing pre-eclampsia before 34 weeks of pregnancy | Before 34 weeks of pregnancy
  YES/NO
Presence of phosphorylation in histone H3 in pregnant women developing pre-eclampsia after 34 weeks of pregnancy | 34 to 41 weeks of pregnancy
  YES/NO
Presence of phosphorylation in histone H4 in pregnant women developing pre-eclampsia before 34 weeks of pregnancy | Before 34 weeks of pregnancy
  YES/NO
Presence of phosphorylation in histone H4 in pregnant women developing pre-eclampsia after 34 weeks of pregnancy | 34 to 41 weeks of pregnancy
  YES/NO
Presence of ubiquitination in histone H2A in pregnant women developing pre-eclampsia before 34 weeks of pregnancy | Before 34 weeks of pregnancy
  YES/NO
Presence of ubiquitination in histone H2A in pregnant women developing pre-eclampsia after 34 weeks of pregnancy | 34 to 41 weeks of pregnancy
  YES/NO
Presence of ubiquitination in histone H2B in pregnant women developing pre-eclampsia before 34 weeks of pregnancy | Before 34 weeks of pregnancy
  YES/NO
Presence of ubiquitination in histone H2B in pregnant women developing pre-eclampsia after 34 weeks of pregnancy | 34 to 41 weeks of pregnancy
  YES/NO
Presence of ubiquitination in histone H3 in pregnant women developing pre-eclampsia before 34 weeks of pregnancy | Before 34 weeks of pregnancy
  YES/NO
Presence of ubiquitination in histone H3 in pregnant women developing pre-eclampsia after 34 weeks of pregnancy | 34 to 41 weeks of pregnancy
  YES/NO
Presence of ubiquitination in histone H4 in pregnant women developing pre-eclampsia before 34 weeks of pregnancy | Before 34 weeks of pregnancy
  YES/NO
Presence of ubiquitination in histone H4 in pregnant women developing pre-eclampsia after 34 weeks of pregnancy | 34 to 41 weeks of pregnancy
  YES/NO
Presence of citrullination in histone H2A in pregnant women developing pre-eclampsia before 34 weeks of pregnancy | Before 34 weeks of pregnancy
  YES/NO
Presence of citrullination in histone H2A in pregnant women developing pre-eclampsia after 34 weeks of pregnancy | 34 to 41 weeks of pregnancy
  YES/NO
Presence of citrullination in histone H2B in pregnant women developing pre-eclampsia before 34 weeks of pregnancy | Before 34 weeks of pregnancy
  YES/NO
Presence of citrullination in histone H2B in pregnant women developing pre-eclampsia after 34 weeks of pregnancy | 34 to 41 weeks of pregnancy
  YES/NO
Presence of citrullination in histone H3 in pregnant women developing pre-eclampsia before 34 weeks of pregnancy | Before 34 weeks of pregnancy
  YES/NO
Presence of citrullination in histone H3 in pregnant women developing pre-eclampsia after 34 weeks of pregnancy | 34 to 41 weeks of pregnancy
  YES/NO
Presence of citrullination in histone H4 in pregnant women developing pre-eclampsia before 34 weeks of pregnancy | Before 34 weeks of pregnancy
  YES/NO
Presence of citrullination in histone H4 in pregnant women developing pre-eclampsia after 34 weeks of pregnancy | 34 to 41 weeks of pregnancy
  YES/NO
Intensity of methylation in histone H2A in pregnant women developing pre-eclampsia before 34 weeks of pregnancy | Before 34 weeks of pregnancy
  Mass spectrometry, quantitative
Intensity of methylation in histone H2A in pregnant women developing pre-eclampsia after 34 weeks of pregnancy | 34 to 41 weeks of pregnancy
  Mass spectrometry, quantitative
Intensity of methylation in histone H2B in pregnant women developing pre-eclampsia before 34 weeks of pregnancy | Before 34 weeks of pregnancy
  Mass spectrometry, quantitative
Intensity of methylation in histone H2B in pregnant women developing pre-eclampsia after 34 weeks of pregnancy | 34 to 41 weeks of pregnancy
  Mass spectrometry, quantitative
Intensity of methylation in histone H3 in pregnant women developing pre-eclampsia before 34 weeks of pregnancy | Before 34 weeks of pregnancy
  Mass spectrometry, quantitative
Intensity of methylation in histone H3 in pregnant women developing pre-eclampsia after 34 weeks of pregnancy | 34 to 41 weeks of pregnancy
  Mass spectrometry, quantitative
Intensity of methylation in histone H4 in pregnant women developing pre-eclampsia before 34 weeks of pregnancy | Before 34 weeks of pregnancy
  Mass spectrometry, quantitative
Intensity of methylation in histone H4 in pregnant women developing pre-eclampsia after 34 weeks of pregnancy | 34 to 41 weeks of pregnancy
  Mass spectrometry, quantitative
Intensity of acetylation in histone H2A in pregnant women developing pre-eclampsia before 34 weeks of pregnancy | Before 34 weeks of pregnancy
  Mass spectrometry, quantitative
Intensity of acetylation in histone H2A in pregnant women developing pre-eclampsia after 34 weeks of pregnancy | 34 to 41 weeks of pregnancy
  Mass spectrometry, quantitative
Intensity of acetylation in histone H2B in pregnant women developing pre-eclampsia before 34 weeks of pregnancy | Before 34 weeks of pregnancy
  Mass spectrometry, quantitative
Intensity of acetylation in histone H2B in pregnant women developing pre-eclampsia after 34 weeks of pregnancy | 34 to 41 weeks of pregnancy
  Mass spectrometry, quantitative
Intensity of acetylation in histone H3 in pregnant women developing pre-eclampsia before 34 weeks of pregnancy | Before 34 weeks of pregnancy
  Mass spectrometry, quantitative
Intensity of acetylation in histone H3 in pregnant women developing pre-eclampsia after 34 weeks of pregnancy | 34 to 41 weeks of pregnancy
  Mass spectrometry, quantitative
Intensity of acetylation in histone H4 in pregnant women developing pre-eclampsia before 34 weeks of pregnancy | Before 34 weeks of pregnancy
  Mass spectrometry, quantitative
Intensity of acetylation in histone H4 in pregnant women developing pre-eclampsia after 34 weeks of pregnancy | 34 to 41 weeks of pregnancy
  Mass spectrometry, quantitative
Intensity of phosphorylation in histone H2A in pregnant women developing pre-eclampsia before 34 weeks of pregnancy | Before 34 weeks of pregnancy
  Mass spectrometry, quantitative
Intensity of phosphorylation in histone H2A in pregnant women developing pre-eclampsia after 34 weeks of pregnancy | 34 to 41 weeks of pregnancy
  Mass spectrometry, quantitative
Intensity of phosphorylation in histone H2B in pregnant women developing pre-eclampsia before 34 weeks of pregnancy | Before 34 weeks of pregnancy
  Mass spectrometry, quantitative
Intensity of phosphorylation in histone H2B in pregnant women developing pre-eclampsia after 34 weeks of pregnancy | 34 to 41 weeks of pregnancy
  Mass spectrometry, quantitative
Intensity of phosphorylation in histone H3 in pregnant women developing pre-eclampsia before 34 weeks of pregnancy | Before 34 weeks of pregnancy
  Mass spectrometry, quantitative
Intensity of phosphorylation in histone H3 in pregnant women developing pre-eclampsia after 34 weeks of pregnancy | 34 to 41 weeks of pregnancy
  Mass spectrometry, quantitative
Intensity of phosphorylation in histone H4 in pregnant women developing pre-eclampsia before 34 weeks of pregnancy | Before 34 weeks of pregnancy
  Mass spectrometry, quantitative
Intensity of phosphorylation in histone H4 in pregnant women developing pre-eclampsia after 34 weeks of pregnancy | 34 to 41 weeks of pregnancy
  Mass spectrometry, quantitative
Intensity of ubiquitination in histone H2A in pregnant women developing pre-eclampsia before 34 weeks of pregnancy | Before 34 weeks of pregnancy
  Mass spectrometry, quantitative
Intensity of ubiquitination in histone H2A in pregnant women developing pre-eclampsia after 34 weeks of pregnancy | 34 to 41 weeks of pregnancy
  Mass spectrometry, quantitative
Intensity of ubiquitination in histone H2B in pregnant women developing pre-eclampsia before 34 weeks of pregnancy | Before 34 weeks of pregnancy
  Mass spectrometry, quantitative
Intensity of ubiquitination in histone H2B in pregnant women developing pre-eclampsia after 34 weeks of pregnancy | 34 to 41 of pregnancy
  Mass spectrometry, quantitative
Intensity of ubiquitination in histone H3 in pregnant women developing pre-eclampsia before 34 weeks of pregnancy | Before 34 weeks of pregnancy
  Mass spectrometry, quantitative
Intensity of ubiquitination in histone H3 in pregnant women developing pre-eclampsia after 34 weeks of pregnancy | 34 to 41 weeks of pregnancy
  Mass spectrometry, quantitative
Intensity of ubiquitination in histone H4 in pregnant women developing pre-eclampsia before 34 weeks of pregnancy | Before 34 weeks of pregnancy
  Mass spectrometry, quantitative
Intensity of ubiquitination in histone H4 in pregnant women developing pre-eclampsia after 34 weeks of pregnancy | 34 to 41 weeks of pregnancy
  Mass spectrometry, quantitative
Intensity of citrullination in histone H2A in pregnant women developing pre-eclampsia before 34 weeks of pregnancy | Before 34 weeks of pregnancy
  Mass spectrometry, quantitative
Intensity of citrullination in histone H2A in pregnant women developing pre-eclampsia after 34 weeks of pregnancy | 34 to 41 weeks of pregnancy
  Mass spectrometry, quantitative
Intensity of citrullination in histone H2B in pregnant women developing pre-eclampsia before 34 weeks of pregnancy | Before 34 weeks of pregnancy
  Mass spectrometry, quantitative
Intensity of citrullination in histone H2B in pregnant women developing pre-eclampsia after 34 weeks of pregnancy | 34 to 41 weeks of pregnancy
  Mass spectrometry, quantitative
Intensity of citrullination in histone H3 in pregnant women developing pre-eclampsia before 34 weeks of pregnancy | Before 34 weeks of pregnancy
  Mass spectrometry, quantitative
Intensity of citrullination in histone H3 in pregnant women developing pre-eclampsia after 34 weeks of pregnancy | 34 to 41 weeks of pregnancy
  Mass spectrometry, quantitative
Intensity of citrullination in histone H4 in pregnant women developing pre-eclampsia before 34 weeks of pregnancy | Before 34 weeks of pregnancy
  Mass spectrometry, quantitative
Intensity of citrullination in histone H4 in pregnant women developing pre-eclampsia after 34 weeks of pregnancy | 34 to 41 weeks of pregnancy
  Mass spectrometry, quantitative
Modifications in histones H2A, H2B, H3 and H4 in women developing pre-eclampsia early on compared with modifications in histones H2A, H2B, H3 and H4 in women with normal pregnancies. | Before 34 weeks of pregnancy
  The presence of methylation, acetylation, phosphorylation, ubiquitination and citrullination in each histone in women developing pre-eclampsia early on will be recorded as YES/NO.
Modifications in histones H2A, H2B, H3 and H4 in women developing pre-eclampsia later on compared with modifications in histones H2A, H2B, H3 and H4 in women with normal pregnancies. | 34 to 41 weeks of pregnancy
  The presence of methylation, acetylation, phosphorylation, ubiquitination and citrullination in each histone in women developing pre-eclampsia later on will be recorded as YES/NO.
Intensity of modifications in histones H2A, H2B, H3 and H4 in women developing pre-eclampsia early on compared with modifications in histones H2A, H2B, H3 and H4 in women with normal pregnancies. | Before 34 weeks of pregnancy
  Mass spectrometry, quantitative
Intensity of modifications in histones H2A, H2B, H3 and H4 in women developing pre-eclampsia later on compared with modifications in histones H2A, H2B, H3 and H4 in women with normal pregnancies. | 34 to 41 weeks of pregnancy
  Mass spectrometry, quantitative

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie BOUVIER, Dr., Principal Investigator — Nîmes University Hospital
Locations (1):
- Nîmes University Hospital, Nîmes, Gard, France

IPD SHARING:
Plan to Share IPD: Undecided
All data collection and management will be carried out by the BESPIM (Biostatistique, Epidémiologie clinique, Santé Publique & Innovation en Méthodologie).
  The conditions of transfer of all or part of the research database are decided by the principal investigator and the research sponsor and are the subject of a written contract.